CLINICAL TRIAL: NCT01559090
Title: A Phase 2, Multicenter, Open-label, Dose-escalation Study to Evaluate the Safety and Tolerability of Intravenous Dose of MEDI-546, a Human Monoclonal Antibody Directed Against Type I Interferon Receptor (IFNAR), in Japanese Subjects With Active Systemic Lupus Erythematosus (SLE).
Brief Title: Safety and Tolerability of Intravenous Dose of MEDI-546 in Japanese Subjects With Systemic Lupus Erythematosus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3461C00002
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Japan; Phase2; Safety; Tolerability; Systemic Lupus Erythematosus; SLE, MEDI-546
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MEDI-546 100 mg IV
  Interventions: Drug: MEDI-546
- 2 (Experimental): MEDI-546 300 mg IV
  Interventions: Drug: MEDI-546
- 3 (Experimental): MEDI-546 1000 mg IV
  Interventions: Drug: MEDI-546

INTERVENTIONS:
Drug: MEDI-546 — Stage I: 100 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 300 mg IV, multiple doses once every 4 wks for 156 wks
  Arms: 1
Drug: MEDI-546 — Stage I: 300 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 300 mg IV, multiple doses once every 4 wks for 156 wks
  Arms: 2
Drug: MEDI-546 — Stage I: 1000 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 1000 mg IV, multiple doses once every 4 wks for 156 wks, the dose at Stage II was changed to 300 mg IV.
  Arms: 3

SUMMARY:
The purpose of this study is to assess safety, tolerability, pharmacokinetics and pharmacodynamics of MEDI-546 in Japanese SLE patients.

DETAILED DESCRIPTION:
A phase 2, multicenter, open-label, dose-escalation study to evaluate the safety and tolerability of intravenous dose of MEDI-546, a human monoclonal antibody directed against type I interferon receptor (IFNAR), in Japanese subjects with active systemic lupus erythematosus (SLE)

ELIGIBILITY:
Inclusion Criteria:

* Fulfils at least 4 of the 11 American College of Rheumatology (ACR) classification criteria for SLE.
* Weight greater than or equal to 40.0 kg.
* Diagnosis of pediatric or adult SLE with chronic disease activity requiring ongoing treatment or observation for ≥ 24 weeks prior to screening.
* Currently receiving stable dose of oral prednisone and/or antimalarials/immunosuppressives.
* Active moderate to severe SLE disease based on SLE disease activity score.

Exclusion Criteria:

* Active severe or unstable neuropsychiatric SLE.
* Active severe SLE-driven renal disease or unstable renal disease.
* Clinically significant active infection including ongoing and chronic infections.
* Known history of a primary immunodeficiency or an underlying condition such as human immunodeficiency virus infection or splenectomy that predisposes the subject to infection.
* Confirmed positive tests for hepatitis B or positive test for hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-04-20 (Actual); Primary Completion 2014-08-19 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Weiss, MD, Study Director — MedImmune LLC
Locations (6):
- Japan (6):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Ōta-ku
  - Research Site, Sendai
  - Research Site, Shimotsuke-shi
  - Research Site, Shinjuku-ku

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDI-546 100 mg IV: Stage I: 100 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 300 mg IV, multiple doses once every 4 wks for 156 wks
- MEDI-546 300 mg IV: Stage I: 300 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 300 mg IV, multiple doses once every 4 wks for 156 wks
- MEDI-546 1000 mg IV: Stage I: 1000 mg IV, single dose and multiple doses once every 4 wks for 48 wks Stage II: 1000 mg IV, multiple doses once every 4 wks for 156 wks, the dose at Stage II was changed to 300 mg IV
Period: Stage I
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Started | 6 | 5 | 6
Completed | 4 | 3 | 3
Not Completed | 2 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 3
Period: Stage II
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Started | 4 | 3 | 2 (One subject who completed Stage I did not agree to participate in Stage II)
Completed | 3 | 3 | 2
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV | Total
Number analyzed (Participants) | 6 | 5 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (12) | 34 (11) | 37 (10) | 38 (11)
Sex/Gender, Customized [Number; unit: male/female]
  Male | 0 | 1 | 0 | 16
  Female | 6 | 4 | 6 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Pharmacokinetic Parameters of MEDI-546 After Single Dose: Cmax
Time Frame: Pre-dose and within 30 minutes after end of infusion on Day 1, Days 2, 8, 15, and 22, and pre-dose on Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Number analyzed (Participants) | 6 | 5 | 6
ug/mL | 41.1 (27.6) | 75.1 (12.5) | 254.8 (20.7)

2. Primary Outcome: Overall Summary of Adverse Events
Time Frame: Stage I (up to 48 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Number analyzed (Participants) | 6 | 5 | 6
Participants
  Any AE | 6 | 5 | 6
  Any AE of grade 3 or higher | 1 | 1 | 1
  Any AE with outcome=death | 0 | 0 | 0
  Any SAE | 2 | 2 | 3
  Any AE leading to discontinuation of IP | 2 | 1 | 1
  Any causally related AE | 5 | 4 | 4
  Any other significant AE | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Parameters of MEDI-546 After Single Dose: AUClast
Time Frame: Pre-dose and within 30 minutes after end of infusion on Day 1, Days 2, 8, 15, and 22, and pre-dose on Day 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug.day/mL
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Number analyzed (Participants) | 6 | 5 | 6
ug.day/mL | 221.5 (18.8) | 666.5 (36.8) | 3151.9 (14.6)

4. Secondary Outcome: Anti-drug Antibody (ADA)
Description: MEDI-546 antibody detection measured by electrochemiluminescence (ECL).
Time Frame: Stage I (up to Week 48)
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
Number analyzed (Participants) | 6 | 5 | 6
Participants
  Positive | 1 | 1 | 1
  Negative | 5 | 4 | 5

ADVERSE EVENTS:
Time Frame: Stage I: 337 to 422 days
Arm/Group | MEDI-546 100 mg IV | MEDI-546 300 mg IV | MEDI-546 1000 mg IV
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/5 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MEDI-546 100 mg IV (N=6) | MEDI-546 300 mg IV (N=5) | MEDI-546 1000 mg IV (N=6)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MEDI-546 100 mg IV (N=6) | MEDI-546 300 mg IV (N=5) | MEDI-546 1000 mg IV (N=6)
Nsopharyngitis (Infections and infestations) | 3 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No